CLINICAL TRIAL: NCT04886882
Title: The Effect of Topical Agents in Cream Formations Containing Magnesium Sulfate on Wound Healing in the Rat Model
Brief Title: Topical Agents Containing Magnesium Sulfate & Wound Healing in the Rat Model
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Istanbul Kent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SakuraDermatology1
Record Dates: First submitted 2021-04-13; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Wound Heal
Keywords: magnesium sulphate; wound healing rat model; hydroxyproline
MeSH Terms: interventions — Centella asiatica extract

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group placebo (Placebo Comparator): Isotonic solution will be administered daily to 6 female rats.
  Interventions: Other: placebo comparator
- Group sham (Sham Comparator): Base cream to be applied twice a day to 6 female rats.
  Interventions: Other: sham comparator
- Group %1 mgso4 (Experimental): Cream containing 1% MgSO4 will be applied twice a day to 6 female rats.
  Interventions: Other: Experimental drug 1
- Group %10 MgSO4 (Experimental): Cream containing 10% MgSO4 will be applied twice a day to 6 female rats.
  Interventions: Other: Experimental drug 2
- Group positive control (Active Comparator): Cream containing centella asiatica will be applied twice a day to 6 female rats.
  Interventions: Drug: Centella asiatica

INTERVENTIONS:
Other: placebo comparator — solution containing 0.9 % sodium chlorine
  Arms: Group placebo
Other: sham comparator — vaseline, beeswax,polyglyceryl-3 diisostearate, sorbitan caprylate, propandiol,benzoic acid, glycerin, water
  Arms: Group sham
Other: Experimental drug 1 — A cream containing 10 % MgSO4.vaseline, beeswaxpolyglyceryl-3 diisostearate, sorbitan caprylate, propandiol,benzoic acid, glycerin, water
  Arms: Group %1 mgso4
Other: Experimental drug 2 — A cream containing 10 % MgSO4.vaseline, beeswax,polyglyceryl-3 diisostearate, sorbitan caprylate, propandiol,benzoic acid, glycerin, water
  Arms: Group %10 MgSO4
Drug: Centella asiatica — A cream containing Centella asiatica
  Arms: Group positive control

SUMMARY:
An experimental study examining wound healing in 5 different groups on 30 rats.

DETAILED DESCRIPTION:
Magnesium topically increases collagen synthesis and angiogenesis, providing faster and higher quality wound healing. In addition, with its analgesic effect, it will also eliminate the pain sensation caused by the wound and increase the quality of life of the patient whose skin integrity is impaired.

ELIGIBILITY:
Inclusion Criteria:

* healthy rats between ages of 8- 12 weeks

Exclusion Criteria:

* weight loss of more than 15% of body weight

Ages: 8 Weeks to 12 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
7th day evaluation | 7th day
  Histopathological evaluation of wound healing comparing with the rate of vascular endothelial growth factor (VEGF), transforming growth factor (TGF-beta) and hydroxyproline at immunohistochemical staining with biopsy on the 7th day.

SECONDARY OUTCOMES:
15th day evaluation | 15th day
  Histopathological evaluation of wound healing comparing with the rate of VEGF, TGF-beta and hydroxyproline at immunohistochemical staining with biopsy on the 15th day.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Hospital, Istanbul, Turkey (Türkiye)